CLINICAL TRIAL: NCT04414514
Title: Exploratory Trial of Ruxolitinib 1.5% Cream for the Treatment of Early Stage Hidradenitis Suppurativa
Brief Title: Topical Ruxolitinib 1.5% for Hidradenitis Suppurativa Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Andrea Zaenglein, Principal Investigator, Professor of Dermatology, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label (Experimental): Topical Ruxolitinib 1.5% Cream, twice daily for 16 weeks
  Interventions: Drug: Ruxolitinib 1.5% Cream

INTERVENTIONS:
Drug: Ruxolitinib 1.5% Cream — Topical Ruxolitinib 1.5% Cream

SUMMARY:
Investigators hypothesize that ruxolitinib 1.5% cream is an effective therapy for HS participants through inhibition of inflammatory activity.

Investigators aim to:

* Demonstrate the clinical efficacy of ruxolitinib 1.5% cream in decreasing the clinical disease activity after 16 weeks of treatment.
* Investigate the impact of ruxolitinib 1.5% cream on skin inflammation through translational analyses of skin biopsy samples.

DETAILED DESCRIPTION:
The primary efficacy measure is the proportion of participants that achieve HiSCR at Week 16 with topical ruxolitinib 1.5% cream as compared to Week 0. The HiSCR is defined as an at least a 50% reduction in the total abscess and inflammatory nodule count (AN count) for all study body sites with no increase in abscess count and no increase in draining fistula count relative to Baseline. The primary efficacy analysis will be carried out on all participants who complete 16 weeks of treatment.

The research study consists of an 8 week screening with 16 weeks open-label portion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age 12 years or older
2. Hidradenitis suppurativa, and should be Hurley Stage I or II, defined as papules, nodules, and/or abscess formation, single or multiple, with or without sinus tracts;
3. Subjects must have a diagnosis of HS for at least 3 months (90 days) prior to Baseline;
4. Active HS lesions must be present in at least one distinct anatomic area;
5. Subject must have at least 3 total inflammatory lesions at the Baseline visit;
6. Subjects who had surgery in the treatment area, should be at least 3 months status post the procedure (this applies to deroofing/marsupialization or excision, not incision & drainage)
7. Subject has a negative TB screening assessment (including a PPD test and/or Quantiferon-TB Gold test equivalent) OR for patients with treated latent TB or negative chest x-ray (CXR posterior-anterior [PA] and lateral view within prior 90 days) at Screening with documentation of treated latent tuberculosis (90 days of treatment).
8. Medications can be continued if they have been at a stable dose for the requisite duration and the dose is not increased during the study period:

   * Biologic medication (such as TNF, IL-12/23 or IL-17 inhibitors): Up to 30% of enrolled participants will be allowed to remain on a concurrent biologic at stable dosage if treated with a stable dose and frequency for 6 months or longer;
   * Oral antibiotic must be a stable dose and frequency for 28 days or longer;
   * Hormone-based therapy (birth control pills or spironolactone) must be a stable dose and frequency for 4 months or longer;
   * Oral retinoids must be on a stable dose and frequency for 90 days or longer;
   * Other topical therapy must be discontinued 14 days prior to the Baseline visit.
   * Child bearing potential: In addition, you must be willing to use a method of contraception during the study period and for 4 weeks after the last dose of study drug. (Note: Periodic abstinence calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable as abstinence.)

Exclusion Criteria:

1. Infection(s) unrelated to HS requiring treatment with:

   * intravenous (IV) anti-infectives (antibiotics, antivirals, antifungals) within 30 days prior to Baseline or;
   * oral anti-infectives (antibiotics, antivirals, antifungals) within 14 days prior to Baseline, except as required as part of an anti-TB regimen;
2. Subject previously treated with a biologic medication but stopped due to lack of effect/sufficient effect as deemed by the investigator.
3. Any other active skin disease or condition (e.g., bacterial, fungal or viral infection) that may interfere with assessment of HS;
4. Pregnant (or considering becoming pregnant) or lactating females Note: Non child bearing potential is defined as surgically sterile with a hysterectomy and/or bilateral oophorectomy OR postmenopausal (defined as amenorrhea at least 12 months before screening, confirmed by FSH levels at screening).
5. Clinically significant abnormal screening laboratory results as evaluated by the Investigator.
6. Subject does not have reliable internet access for weekly electronic surveys;
7. Subject is considered by the Study Investigator, for any reason, to be an unsuitable candidate for the study.
8. Excluded prohibited concomitant medication and procedures include: JAK inhibitors (systemic or topical (eg, ruxolitinib, tofacitinib, baricitinib, filgotinib, lestaurtinib, and pacritinib) within 4 weeks of Screening ; surgical, laser, or IPL intervention in area with HS lesion within 3 months of Screening, except for rescue lesional treatment; systemic corticosteroid within 4 weeks; use of topical creams, ointments, gels, and liquids except the study therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
HiSCR | The primary efficacy analysis will be carried out on all participants who complete 16 weeks of treatment.
  The HiSCR is defined as at least a 50% reduction in the total abscess and inflammatory nodule count (AN count) for all study body sites with no increase in abscess count and no increase in draining fistula count relative to Baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided